CLINICAL TRIAL: NCT04336956
Title: Covid-19 Pediatric Observatory
Acronym: PANDOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other); Groupe de Pathologies Infectieuses Pédiatriques (GPIP) (Other); Société Française de Pédiatrie (Unknown); Francophone Pediatric Resuscitation and Emergency Group (GFRUP) (Other)
Responsible Party: Sponsor
Other Study IDs: PANDOR
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: children; pediatric department
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospitalized children with Covid19: - Children < 18 years old Patients under 18 years old, admitted in French pediatric wards with a confirmed COVID-19 infection on Nasal and pharyngeal swab specimens or blood samples tested positive for 2019-nCoV nucleic acid using real-time reverse-transcriptase polymerase-chain-reaction (RT- PCR) assay; or on typical chest CT signs
  Interventions: Other: hospitalized children with Covid19

INTERVENTIONS:
Other: hospitalized children with Covid19 — All patients under 18 years hospitalized with a covid19 diagnosis

SUMMARY:
In early December 2019, cases of pneumonia of unknown origin were reported in Wuhan, Hubei Province in the People's Republic of China. The disease spreads rapidly and the number of sick people is increasing. On January 3, 2020 a new virus of the coronavirus family is identified in samples of bronchoalveolar lavage fluid from a patient in Wuhan and subsequently confirmed as the cause of these pneumonias. On 7 January 2020, the World Health Organization (WHO) designated it as the new coronavirus 2019 (i.e. 2019-nCoV). On 11 February 2020, the WHO designated the disease associated with 2019-nCoV as coronavirus 2019 disease (COVID-19). On 12 March, WHO announced that the COVID-19 outbreak is a pandemic.

As of March 24, 2020, more than 375,000 cases of COVID-19 had been diagnosed with more than 16,000 deaths attributed to this virus. (Ref WHO https://www.who.int/emergencies/diseases/novel-coronavirus-2019 ).

In France, the number of cases rose from 105 cases at the end of February to 19615 confirmed cases on March 24. (Source Public Health France). Most of the cases are adults. However, children are not completely spared and serious cases have been described. These severe cases can be respiratory or extra-respiratory (e.g. myocarditis). We also know that pediatric and adult cases differ in terms of clinical, biological and imaging findings, particularly chest CT scans. However, the description of paediatric pictures, especially severe forms and the involvement of children suffering from co-morbidities, remains poorly reported. Finally, the risk factors for serious cases in children remain largely unknown.

This observatory aim to describe the clinical phenotypes of hospitalized pediatric patients with Covid19 in France, according to age groups. Moreover for a subgroup of patients, informations regarding the long covid will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Children < 18 years old
* Admitted in French pediatric wards
* With a confirmed COVID-19 infection. ( on Nasal and pharyngeal swab specimens or blood samples tested positive for 2019-nCoV nucleic acid using real-time reverse-transcriptase polymerase-chain-reaction (RT- PCR) assay; or on typical chest CT signs

Exclusion Criteria:

* Expressed refusal to participate

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children hospitalized with covid19
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of children with severe or critical form. | Day 14

SECONDARY OUTCOMES:
Percentage of children requiring intensive care support | at admission
Percentage of children requiring intensive care support | at day 14
Clinical symptoms of children | at admission
  requiring intensive care support or not
Clinical symptoms of children | day 14
  requiring intensive care support or not
Biological results of children | at admission
  requiring intensive care support or not
Biological results of children | day 14
  requiring intensive care support or not
CT chest of children | at admission
  requiring intensive care support or not
Pulmonary echography | Day 14
  requiring intensive care support or not
nasopharynx SARScov2 PCR | at admission
nasopharynx sarscov2 load | at day 7
  if available
nasopharynx multiplex PCR | at admission
  if available
number of hospital days | up to 12months
  days
Evaluation of long covid | up to 12months

CONTACTS AND LOCATIONS:
Locations (76):
- France (76):
  - Chu Felix Guyon, Saint-Denis, La Réunion
  - Ch St Esprit, Agen
  - Ch General Aix En Provence -, Aix-en-Provence
  - CHU Angers, Angers
  - CH d'ANGOULEME, Angoulème
  - Pringy - Ch D'Annecy, Annecy
  - CH Argenteuil, Argenteuil
  - Ch Armentieres, Armentières
  - CH Arpajon, Arpajon
  - Ch Auxerre, Auxerre
  - CH GENERAL Henri Duffaut, Avignon
  - CHU de BESANCON, Besançon
  - Hopital Femme Enfant, Caen
  - Ch de Pontoise, Cergy-Pontoise
  - Ch W. Morey, Chalon-sur-Saône
  - CH de CHAMBERY, Chambéry
  - Ch Hotel Dieu, Chartres
  - CHU Estaing, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Hopital Louis Mourrier, Colombes
  - CH Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier intercommunal de Creteil, Créteil
  - Ch de Dax, Dax
  - Hopital D'Enfants Chu Dijon, Dijon
  - CH Louviers Val de Reuil, Elbeuf
  - CH Jean Monnet, Épinal
  - CH Gonesse, Gonesse
  - CH d'HYERES, Hyères
  - Ch de Marne La Vallee, Jossigny
  - Chru de Grenoble, La Tronche
  - CHGénéral du HAVRE, Le Havre
  - Hopital Jeanne de Flandre, Lille
  - Hopital Roger Salengro - Lille, Lille
  - Hopital Saint Vincent de Paul, Lille
  - Ch de Longjumeau, Longjumeau
  - Lorient - Ch de Bretagne Sud, Lorient
  - Hopital Femme Mere Enfant-Bron, Lyon
  - Hopital de Mantes, Mantes-la-Jolie
  - Hopital Nord Enfants, Marseille
  - Hopital de Meaux, Meaux
  - Ch de Melun, Meulin
  - CH de Montargis, Montargis
  - CH de MONTBRISON, Montbrison
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHRU de Nancy, Nancy
  - Nantes - Hopital Mere Enfant, Nantes
  - Ch de Neuilly Sur Seine, Neuilly-sur-Seine
  - Hopital Lenval, Nice
  - CHU Nimes Caremeau, Nîmes
  - Chr Orleans, Orléans
  - Assistance Publique Hôpitaux de Paris, Paris
  - Hopital St Jean Roussillon, Perpignan
  - POISSY - CH de POISSY, Poissy
  - QUIMPER - CH de Cornouaille, Quimper
  - RANG du FLIERS - C.H.A.M., Rang-du-Fliers
  - Hopital Américain CHU REIMS, Reims
  - CH RODEZ, Rodez
  - CH de ROMANS, Romans-sur-Isère
  - Chu Rouen, Rouen
  - Hopital Charles-Nicolle, Rouen
  - Ch de Saint Denis, Saint-Denis
  - Chu St Etienne, Saint-Etienne
  - Ch Du Pays Du Mont Blanc, Sallanches
  - Chg Salon de Provence, Salon-de-Provence
  - Ch de Saint Malo, St-Malo
  - CH Hautepierre, Strasbourg
  - CH Tarbes, Tarbes
  - CH Bel Air, Thionville
  - Hopital Sainte Musse, Toulon
  - CHU Toulouse-hôpital des Enfants, Toulouse
  - Hôpital Gatien De Clocheville, Tours
  - Hôpital Nord Franche-Comté, Trévenans
  - CH de TROYES, Troyes
  - Ch Bretagne Atlantique, Vannes
  - Ch Le Chesnay, Versailles
  - Hopital de Villeneuve Saint Georges, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rybak A, Ouldali N, Werner A, Casha P, Robert B, de Pontual L, Bechet S, Cahn-Sellem F, Angoulvant F, Cohen R, Levy C; PANDOR study group. Characteristics of Children Hospitalized for Acute COVID-19 in France From February 2020 to December 2023. Pediatr Infect Dis J. 2025 Apr 1;44(4):346-350. doi: 10.1097/INF.0000000000004681. Epub 2025 Feb 14. PMID 39961110
- See also: Association of Intravenous Immunoglobulins Plus Methylprednisolone vs Immunoglobulins Alone With Course of Fever in Multisystem Inflammatory Syndrome in Children — https://pubmed.ncbi.nlm.nih.gov/33523115/
- See also: Factors Associated With Severe SARS-CoV-2 Infection — https://pubmed.ncbi.nlm.nih.gov/33323493/
- See also: Educational Setting and SARS-CoV-2 Transmission Among Children With Multisystem Inflammatory Syndrome: A French National Surveillance System — https://pubmed.ncbi.nlm.nih.gov/34765576/
- See also: Analysis of COVID-19 Vaccination Status Among Parents of Hospitalized Children Younger Than 5 Years With SARS-CoV-2 Infection During the Delta and Omicron Waves — https://pubmed.ncbi.nlm.nih.gov/36383384/